CLINICAL TRIAL: NCT00875004
Title: Research Factors Predictive of Treatment Failure With Erythropoietin Beta (NeoRecormon®) in Patients With Solid Tumors Treated With Chemotherapy
Brief Title: Epoetin Beta in Patients Undergoing Chemotherapy for Solid Tumors
Acronym: PLATON
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After two years of trial initiation, only 27 out of 300 patients were included. During this period, the international recommendations for the use of COOL were modified.
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000633325; CLCC-VA-2007/21; CLCC-AFSSAPS-A70755-52; INCA-RECF0639; EUDRACT-2007-003615-31; ROCHE-CLCC-PLATON
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2024-06-26 (Actual); Status verified 2022-08

CONDITIONS: Anemia; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: anemia; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Anemia | interventions — epoetin beta; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Erythropoietin beta (Experimental)
  Interventions: Biological: epoetin beta; Drug: systemic chemotherapy; Procedure: quality-of-life assessment

INTERVENTIONS:
Biological: epoetin beta
Drug: systemic chemotherapy
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Epoetin beta may cause the body to make more red blood cells and may prevent or reduce side effects in patients undergoing chemotherapy for solid tumors.

PURPOSE: This clinical trial is studying how well epoetin beta works in patients undergoing chemotherapy for solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Identify factors predictive of treatment failure in patients with solid tumors treated with epoetin beta while undergoing chemotherapy.

Secondary

* Evaluate the impact of achieving target hemoglobin levels (i.e., hemoglobin > 11 g/dL) after 8 weeks of treatment with epoetin beta.
* Evaluate changes in hemoglobin levels from baseline to after 8 weeks of treatment with epoetin beta.
* Evaluate the tolerability of epoetin beta in these patients.
* Evaluate the quality of life of these patients.

OUTLINE: This is a multicenter study.

Patients receive epoetin beta subcutaneously once a week for ≥ 8 weeks in the absence of disease progression or unacceptable toxicity.

Patients complete a quality-of-life questionnaire (FACT-An) at baseline and after 8 weeks of treatment.

ELIGIBILITY:
Inclusion criteria :

* Age > 18 years
* Hemoglobin levels between [ > 9g/dl - < 11 g/dl ] .
* Patient requiring erythropoietine beta treatment for a foreseeable duration of at least 8 weeks under the same chemotherapy protocol.
* Patient with cancer undergoing chemotherapy
* Patient without EPO within 6 months prior to current chemotherapy.
* WHO 2 performance status (Appendix 1).
* Patient information and signature of informed consent or legal representative

Exclusion criteria :

* Hemoglobin < 9 g/dl or > 11 g/dl
* Patient with cancer not treated with chemotherapy (targeted therapy, hormone therapy, etc…)
* Patient with cancer treated with concomitant radiation chemotherapy.
* Co-treated with Epo beta and scheduled transfusion prior to inclusion.
* Hypersensitivity to the active substance or one of the NeoRecormon excipients®
* Poorly controlled high blood pressure
* Pregnant woman, likely to be pregnant or breastfeeding,
* Persons deprived of liberty or under guardianship,
* Unable to undergo medical follow-up for geographic, social or psychological reasons.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-12-07 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2011-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment failure (changes in hemoglobin levels) | From date of randomization until the week 8
  The 8th week of treatment assessment defines the patient on erythropoeitine beta (NeoRecormon®) treatment for failure or success

CONTACTS AND LOCATIONS:
Overall Officials: Damien Pouessel, MD, Principal Investigator — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (1):
- Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beguin Y. Prediction of response to treatment with recombinant human erythropoietin in anaemia associated with cancer. Med Oncol. 1998 Aug;15 Suppl 1:S38-46. PMID 9785336
- [Background] Bokemeyer C, Aapro MS, Courdi A, Foubert J, Link H, Osterborg A, Repetto L, Soubeyran P. EORTC guidelines for the use of erythropoietic proteins in anaemic patients with cancer. Eur J Cancer. 2004 Oct;40(15):2201-16. doi: 10.1016/j.ejca.2004.07.015. PMID 15454245
- [Background] Bonomi AE, Cella DF, Hahn EA, Bjordal K, Sperner-Unterweger B, Gangeri L, Bergman B, Willems-Groot J, Hanquet P, Zittoun R. Multilingual translation of the Functional Assessment of Cancer Therapy (FACT) quality of life measurement system. Qual Life Res. 1996 Jun;5(3):309-20. doi: 10.1007/BF00433915. PMID 8763799
- [Background] Cella D. The Functional Assessment of Cancer Therapy-Anemia (FACT-An) Scale: a new tool for the assessment of outcomes in cancer anemia and fatigue. Semin Hematol. 1997 Jul;34(3 Suppl 2):13-9. PMID 9253779
- [Background] Curt GA, Breitbart W, Cella D, Groopman JE, Horning SJ, Itri LM, Johnson DH, Miaskowski C, Scherr SL, Portenoy RK, Vogelzang NJ. Impact of cancer-related fatigue on the lives of patients: new findings from the Fatigue Coalition. Oncologist. 2000;5(5):353-60. doi: 10.1634/theoncologist.5-5-353. PMID 11040270
- [Background] Del Mastro L, Gennari A, Donati S. Chemotherapy of non-small-cell lung cancer: role of erythropoietin in the management of anemia. Ann Oncol. 1999;10 Suppl 5:S91-4. doi: 10.1093/annonc/10.suppl_5.s91. PMID 10582148
- [Background] Demetri GD, Kris M, Wade J, Degos L, Cella D. Quality-of-life benefit in chemotherapy patients treated with epoetin alfa is independent of disease response or tumor type: results from a prospective community oncology study. Procrit Study Group. J Clin Oncol. 1998 Oct;16(10):3412-25. doi: 10.1200/JCO.1998.16.10.3412. PMID 9779721
- [Background] Glaspy J, Bukowski R, Steinberg D, Taylor C, Tchekmedyian S, Vadhan-Raj S. Impact of therapy with epoetin alfa on clinical outcomes in patients with nonmyeloid malignancies during cancer chemotherapy in community oncology practice. Procrit Study Group. J Clin Oncol. 1997 Mar;15(3):1218-34. doi: 10.1200/JCO.1997.15.3.1218. PMID 9060566
- [Background] Groopman JE, Itri LM. Chemotherapy-induced anemia in adults: incidence and treatment. J Natl Cancer Inst. 1999 Oct 6;91(19):1616-34. doi: 10.1093/jnci/91.19.1616. PMID 10511589
- [Background] Littlewood TJ. The impact of hemoglobin levels on treatment outcomes in patients with cancer. Semin Oncol. 2001 Apr;28(2 Suppl 8):49-53. doi: 10.1016/s0093-7754(01)90213-1. PMID 11395853
- [Background] Bokemeyer C, Aapro MS, Courdi A, Foubert J, Link H, Osterborg A, Repetto L, Soubeyran P; European Organisation for Research and Treatment of Cancer (EORTC) Taskforce for the Elderly. EORTC guidelines for the use of erythropoietic proteins in anaemic patients with cancer: 2006 update. Eur J Cancer. 2007 Jan;43(2):258-70. doi: 10.1016/j.ejca.2006.10.014. Epub 2006 Dec 19. PMID 17182241
- [Background] Aapro M, Coiffier B, Dunst J, Osterborg A, Burger HU. Effect of treatment with epoetin beta on short-term tumour progression and survival in anaemic patients with cancer: A meta-analysis. Br J Cancer. 2006 Dec 4;95(11):1467-73. doi: 10.1038/sj.bjc.6603481. Epub 2006 Nov 21. PMID 17117175
- [Background] Oberhoff C. Speed of haemoglobin response in patients with cancer: a review of the erythropoietic proteins. Support Care Cancer. 2007 Jun;15(6):603-611. doi: 10.1007/s00520-006-0191-x. Epub 2007 Feb 3. PMID 17277926
- [Background] Pujade-Lauraine E, Topham C. Once-weekly treatment of anemia in patients with cancer: a comparative review of epoetins. Oncology. 2005;68(2-3):122-9. doi: 10.1159/000086957. Epub 2005 Jul 7. PMID 16015034
- [Background] Veys N, Dhondt A, Lameire N. Pain at the injection site of subcutaneously administered erythropoietin: phosphate-buffered epoetin alpha compared to citrate-buffered epoetin alpha and epoetin beta. Clin Nephrol. 1998 Jan;49(1):41-4. PMID 9491285
- [Background] Thomas ML. Impact of anemia and fatigue on quality of life in cancer patients: a brief review. Med Oncol. 1998 Aug;15 Suppl 1:S3-7. PMID 9785330
- [Background] Vogelzang NJ, Breitbart W, Cella D, Curt GA, Groopman JE, Horning SJ, Itri LM, Johnson DH, Scherr SL, Portenoy RK. Patient, caregiver, and oncologist perceptions of cancer-related fatigue: results of a tripart assessment survey. The Fatigue Coalition. Semin Hematol. 1997 Jul;34(3 Suppl 2):4-12. PMID 9253778
- [Background] Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage. 1997 Feb;13(2):63-74. doi: 10.1016/s0885-3924(96)00274-6. PMID 9095563
- [Background] Harrell FE Jr, Lee KL, Mark DB. Multivariable prognostic models: issues in developing models, evaluating assumptions and adequacy, and measuring and reducing errors. Stat Med. 1996 Feb 28;15(4):361-87. doi: 10.1002/(SICI)1097-0258(19960229)15:43.0.CO;2-4. PMID 8668867